CLINICAL TRIAL: NCT07094698
Title: The Effects of Sacral Stimulation on Urinary Incontinence, Constipation, Sexual Function, and Daily Living Activities in Women With Low Back Pain
Brief Title: Sacral Stimulation in Women With Low Back Pain: Effects on Pelvic Functions and Daily Life
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Muhammed Fatih Kavak, Dr., Uskudar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 61351342/020-1199
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pelvic Floor Dysfunction; Low Back Pain
Keywords: sacral stimulation; Activities of daily living; sexual function
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Forty female volunteers aged 18 to 65 years with complaints of urinary incontinence will be included. Low-frequency (2-10 Hz) current with a pulse duration of 200 μs will be applied for 30 minutes, 5 days a week, under the supervision of a physiotherapist for 6 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacral stimulation (Experimental): A low-frequency (2-10 Hz) current with a pulse duration of 200 μs will be applied for 30 minutes, 5 days a week, under the supervision of a physiotherapist for 6 weeks.
  Interventions: Other: sacral stimulation

INTERVENTIONS:
Other: sacral stimulation — A low-frequency (2-10 Hz) current with a pulse duration of 200 μs will be applied for 30 minutes, 5 days a week, under the supervision of a physiotherapist for 6 weeks.

SUMMARY:
Pelvic floor dysfunction is a term used to describe a variety of disorders involving moderate to severe impairment of the pelvic floor muscles. The pelvic floor is a layer of muscle designed to support the abdominal organs and maintain urethral, anal, and vaginal continence. It includes the pubococcygeus, puborectalis, and iliococcygeus muscles. Pelvic floor muscle dysfunction, which causes significant morbidity particularly in women, is associated with stress urinary incontinence, anal and fecal incontinence, pelvic organ prolapse, and sexual dysfunction, all of which can negatively affect quality of life in women. Moreover, various comorbid conditions such as back and neck pain, asthma, cardiovascular diseases, and psychiatric disorders are also associated with pelvic floor dysfunction.

In patients diagnosed with lumbar disc herniation, changes in pelvic floor muscle strength have been observed. These changes may be accompanied by urinary and sexual problems. Individuals with low back pain are at twice the risk of urinary incontinence compared to those without back pain, and strengthening of the pelvic floor muscles has been shown to reduce back pain.

This study aims to understand the characteristics of transcutaneous sacral nerve stimulation, examine the neurophysiological basis of this treatment method, and evaluate its potential for future innovative approaches.

DETAILED DESCRIPTION:
Pelvic floor dysfunction is a term used to describe various disorders involving moderate to severe impairment of the pelvic floor muscles. The pelvic floor is a layer of muscle designed to support the abdominal organs and maintain urethral, anal, and vaginal continence. It is collectively referred to as the levator ani and includes the pubococcygeus, puborectalis, and iliococcygeus muscles. Pelvic floor muscle dysfunction, which causes significant morbidity especially in women, is associated with stress urinary incontinence, anal and fecal incontinence, pelvic organ prolapse, and sexual dysfunction. These conditions negatively affect women's quality of life. Additionally, several comorbidities such as back and neck pain, asthma, cardiovascular diseases, and psychiatric disorders are also associated with pelvic floor dysfunction.

In patients diagnosed with lumbar disc herniation, changes in pelvic floor muscle strength have been observed. These changes may be accompanied by urinary and sexual problems. Individuals with low back pain are at twice the risk of developing urinary incontinence compared to those without low back pain. It has been shown that strengthening the pelvic floor muscles can help reduce low back pain.

This study is planned to be conducted at Istanbul Medipol Acıbadem Regional Hospital between May 1, 2025, and December 1, 2025. All participants will be provided with detailed information about the study, and written informed consent will be obtained from those who agree to participate voluntarily.

All individuals included in the study will complete a demographic information form, which includes age, gender, height, weight, medication use, family history, and smoking status.

The study population will consist of 40 voluntary female participants between the ages of 18 and 65 who have complaints of urinary incontinence. All participants will be placed in a single group and will receive a low-frequency (2-10 Hz), 200 μs pulse duration current for 30 minutes a day, 5 days a week for 6 weeks under the supervision of a physiotherapist.

Data collection tools in this study include:

The Sociodemographic Information Form, The Oswestry Low Back Pain Disability Questionnaire to assess low back pain levels, The King's Health Questionnaire (KHQ) to evaluate urinary incontinence, The Constipation Severity Instrument (CSI) to assess constipation, The Sexual Quality of Life Questionnaire - Female (SQoL-F) to evaluate sexual dysfunction.

Necessary permissions have been obtained from the original authors for the use of all questionnaires with established validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

Having complaints of urinary incontinence Having complaints of low back pain Diagnosed with constipation according to Rome IV criteria Women with pelvic floor dysfunction Being under 65 years of age Having normal mood and memory functions Being able to speak Turkish Being literate Voluntarily agreeing to participate in the study

Exclusion Criteria:

Neuromuscular diseases (such as Multiple Sclerosis, Parkinson's disease, Myasthenia Gravis, etc.) Malignant tumors Diabetes and other serious medical conditions Pelvic radiation, rectal surgery, spinal surgery Hysterectomy Pelvic inflammation Urinary tract infection Vaginitis Pacemaker implantation Pregnancy Cognitive impairment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to the nature of the condition being studied, only female participants will be included in the study.
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Severity of constipation | through study completion, an average of 2 months.
  Constipation severity will be measured using the Constipation Severity Instrument (CSI). The scale consists of a total of 16 questions. The CSI includes subscales for colonic inertia, stool obstruction, and pain. The score for the colonic inertia subscale ranges from 0 to 29, the stool obstruction subscale from 0 to 28, and the pain subscale from 0 to 16. Therefore, the total possible score on the CSI ranges from 0 to 73. Higher scores on the scale indicate more severe symptoms.
Severity of urinary incontinence | through study completion, an average of 2 months.
  Urinary incontinence will be assessed using the King's Health Questionnaire (KHQ). The questionnaire, which consists of 32 items divided into two parts, is widely used to evaluate the quality of life in patients with incontinence. In addition to two single-item questions addressing general health status and the impact on quality of life, it includes seven multi-item subscales. These subscales are role limitations, physical limitations, social limitations, personal relationships limitations, emotional problems, sleep and energy disturbances related to incontinence, and severity measures of incontinence.
  The second part consists of an 11-item symptom severity scale that evaluates the presence and severity of urinary symptoms. Scores on the symptom severity scale range from 0 (best) to 30 (worst). Scores for the other KHQ domains range from 0 (best) to 100 (worst).
Sexual quality of life | through study completion, an average of 2 months.
  This scale is a six-point Likert type and consists of 18 items. Each item is expected to be answered based on the respondent's sexual life over the past four weeks. Each item is scored between 1 and 6. The total score on the scale ranges from 18 to 108. A higher score indicates better sexual quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: muhammed fatih kavak, dr, Study Director — Uskudar University
Locations (1):
- Medipol Acıbadem Regional Hospital, Istanbul, Turkey (Türkiye)